CLINICAL TRIAL: NCT05276336
Title: The Effect of Early Radiofrequency Turbinate Reduction, Intranasal Steroid, and Antihistamine H-1 on Persistent Allergic Rhinitis: A Randomized Clinical Trial
Brief Title: The Effect of Early Radiofrequency Turbinate Reduction on Persistent Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nina Irawati, Head of Allergy Immunology Division, Otorhinolaryngology Head and Neck Surgery Department, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-08-0974
Record Dates: First submitted 2022-02-18; First posted 2022-03-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis
Keywords: allergic; histamine antagonist; radiofrequency turbinate reduction; rhinitis; steroid
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects will receive radiofrequency turbinate reduction done in the outpatient clinic, followed by pharmacology treatment (intranasal steroid and AH-1) for 8 weeks.
  Interventions: Procedure: Radiofrequency turbinate reduction; Drug: Pharmacology treatment
- Control Group (Active Comparator): Subjects in the control group will receive only the pharmacology treatment for 8 weeks.
  Interventions: Drug: Pharmacology treatment

INTERVENTIONS:
Procedure: Radiofrequency turbinate reduction — Before the radiofrequency turbinate reduction procedure, local anaesthesia will be given by applying a cotton tamponade soaked in lidocaine adrenaline 1:5000 titration and added with xylocaine gel for 10 minutes in both nostrils. Then, a mixture of 1 mL of lidocaine 2% and 2 mL of sodium chloride 0,9% will be infiltrated to both nostrils using 3 mL and 1 mL needles until the inferior turbinates are pale. The radiofrequency probe (made by Sutter, both in monopolar and bipolar modes) will be inserted to the distal inferior turbinate until the black line from the probe is inside the inferior turbinate (approximately 10-12 mm). The procedure will be done for 10 seconds and the insertion of the probe can be done in 2-3 sites. After this, subjects from this group will be treated with pharmacology treatment using intranasal steroid and AH-1 according to ARIA WHO guideline 2008, similar to the pharmacology treatment received by the control group.
  Arms: Intervention Group
Drug: Pharmacology treatment — Subjects will be treated with intranasal steroid and AH-1 according to ARIA WHO guideline 2008. Fluticasone furoate will be given twice a day with two sprays (100 µg) for each nostril for 2 weeks, then continue for once a day with two sprays (100 µg). Antihistamine H-1 is given 10 mg, once a day. Pharmacology treatment is given for 4 weeks, then intranasal steroid will be continued for another 4 weeks.
  Other Names: Standard treatment

SUMMARY:
The primary outcome of this study is to evaluate the effect of radiofrequency turbinate reduction as an initial treatment on clinical improvement (using visual analogue scale based on total nasal symptoms score, peak nasal inspiratory flow, and turbinate size using ImageJ), inflammatory mediators (ELISA from nasal secretions was performed to measure ECP, IL-5, and HSP-70), and remodeling markers (through nasal biopsy followed by immunohistochemistry examination to evaluate MMP-9, TIMP-1, and PAI-1).

In this randomized, controlled trial, 32 patients with moderate-severe persistent AR were randomly divided into 2 groups. Intervention group received radiofrequency turbinate reduction followed by intranasal steroid and antihistamine H-1(AH-1), control group received intranasal steroid and AH-1. Both groups were evaluated for clinical improvement in week 4 and 8 after treatment, inflammatory mediators and remodeling markers in week 4 after treatment.

DETAILED DESCRIPTION:
The study compares 2 groups of moderate-severe persistent allergic rhinitis (AR). The intervention group receives radiofrequency turbinate reduction followed by pharmacology treatment (intranasal steroid and AH-1) while the control group receives only pharmacology treatment.

Diagnosis of AR will be made through clinical history, physical examination, and skin puncture test. Patients aged 18-55 years old with moderate-severe persistent AR who come to the outpatient clinic and have signed the informed consent form will be included in this study. Moderate-severe AR is defined as having AR symptoms for more than 4 days in a week and more than 4 weeks, with symptoms affecting the subjects' quality of life. Patients will be assigned to two groups of treatment randomly with a single blind block randomization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate-severe persistent allergic rhinitis who come to the outpatient clinic and has signed the informed consent form.

Exclusion Criteria:

* Smokers
* Septum deviation in nasal valve without septal swell body
* Unilateral inferior turbinate hypertrophy caused by septum deviation
* Pregnant
* Severe systemic disease
* Acute rhinitis or rhinosinusitis within 6 weeks before the study period
* Nasal polyp
* Nasal or paranasal tumor
* Subjects who had received other methods of inferior turbinate reduction, posterior nasal neurectomy, functional endoscopic sinus surgery, Caldwell Luc
* Subjects who had received topical steroid for 4 weeks before the study period
* Coagulation disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
VAS score based on TNSS at baseline | Evaluation is done at baseline
  Clinical symptoms was evaluated by visual analogue scale (VAS) based on total nasal symptoms score (TNSS). Total nasal symptoms score are based on four symptoms, which are rhinorrea, sneezing, itchy nose, and nose obstruction. Each symptom will be given a score between 1 (most mild symptom) until 5 (most severe symptom). The minum score for VAS based on TNSS is 4 (most mild symptom) and the maximum score is 40 (most severe symptom). VAS score less than five indicates a controlled rhinitis allergy symptoms, while ≥ 5 indicates that symptoms are not controlled.
VAS score based on TNSS at week 4 | Evaluation is done at week 4
  Clinical symptoms was evaluated by visual analogue scale (VAS) based on total nasal symptoms score (TNSS). Total nasal symptoms score are based on four symptoms, which are rhinorrea, sneezing, itchy nose, and nose obstruction. Each symptom will be given a score between 1 (most mild symptom) until 5 (most severe symptom). The minum score for VAS based on TNSS is 4 (most mild symptom) and the maximum score is 40 (most severe symptom). VAS score less than five indicates a controlled rhinitis allergy symptoms, while ≥ 5 indicates that symptoms are not controlled.
VAS score based on TNSS at week 8 | Evaluation is done at week 8
  Clinical symptoms was evaluated by visual analogue scale (VAS) based on total nasal symptoms score (TNSS). Total nasal symptoms score are based on four symptoms, which are rhinorrea, sneezing, itchy nose, and nose obstruction. Each symptom will be given a score between 1 (most mild symptom) until 5 (most severe symptom). The minum score for VAS based on TNSS is 4 (most mild symptom) and the maximum score is 40 (most severe symptom). VAS score less than five indicates a controlled rhinitis allergy symptoms, while ≥ 5 indicates that symptoms are not controlled.
Size of inferior turbinate at baseline | Evaluation is done at baseline
  The inferior turbinate was evaluated by using nasoendoscopy and Image J™ program was used to determine the size of inferior turbinate.
Size of inferior turbinate at week 4 | Evaluation is done at week 4
  The inferior turbinate was evaluated by using nasoendoscopy and Image J™ program was used to determine the size of inferior turbinate.
Size of inferior turbinate at week 8 | Evaluation is done at week 8
  The inferior turbinate was evaluated by using nasoendoscopy and Image J™ program was used to determine the size of inferior turbinate.
PNIF value at baseline | Evaluation is done at baseline
  Nasal airflow resistance was evaluated using In-Check Nasal Inspiratory Flow Meter by Clement Clarke International Itd England. The examination was repeated for three times with 30 seconds paused and the highest value was taken.
PNIF value at week 4 | Evaluation is done at week 4
  Nasal airflow resistance was evaluated using In-Check Nasal Inspiratory Flow Meter by Clement Clarke International Itd England. The examination was repeated for three times with 30 seconds paused and the highest value was taken.
PNIF value at week 8 | Evaluation is done at week 8
  Nasal airflow resistance was evaluated using In-Check Nasal Inspiratory Flow Meter by Clement Clarke International Itd England. The examination was repeated for three times with 30 seconds paused and the highest value was taken.
Inflammatory mediators at baseline | Evaluation is done at baseline
  Inflammatory mediators that will be evaluated are IL-5, ECP, and HSP-70. They were examined from nasal secretions and enzyme-linked immunosorbent assay (ELISA) spectrophotometry is used to evaluate the amount of IL-5, ECP, and HSP-70 in both groups
Inflammatory mediators at week 4 | Evaluation is done at week 4
  Inflammatory mediators that will be evaluated are IL-5, ECP, and HSP-70. They were examined from nasal secretions and enzyme-linked immunosorbent assay (ELISA) spectrophotometry is used to evaluate the amount of IL-5, ECP, and HSP-70 in both groups
Remodeling components at baseline | Evaluation is done at baseline
  Remodeling components that will be evaluated are MMP-9, TIMP-1, and PAI-1. They will be assessed using immunihistochemistry from tissue biopsy of inferior turbinate.
Remodeling components at week 4 | Evaluation is done at week 4
  Remodeling components that will be evaluated are MMP-9, TIMP-1, and PAI-1. They will be assessed using immunihistochemistry from tissue biopsy of inferior turbinate.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Irawati, MD, Principal Investigator — Indonesia University
Locations (1):
- RSUPN Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia